CLINICAL TRIAL: NCT02691039
Title: N.E.W. Keiki - Nutrition + Exercise + Weight Management Programs: Family-based Intervention to Combat Childhood Obesity in Hawai'i
Brief Title: NEW Keiki Family Based Intervention to Combat Childhood Obesity
Status: Completed | Type: Observational
Sponsor: Malia Shimokawa, MD (Other)
Responsible Party: Sponsor-Investigator, Malia Shimokawa, MD, Medical Director, KMCWC Multidisciplinary Clinics, Hawaii Pacific Health
Organization: Hawaii Pacific Health (Other)
Other Study IDs: 2013-075
Record Dates: First submitted 2014-03-25; First posted 2016-02-25 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to create a database to collect information about the NEW Keiki Program. The information collected for this project will be used to evaluate the program. The NEW Keiki program promotes healthy lifestyles and behavior changes.

DETAILED DESCRIPTION:
A database containing pre and post program information will be developed. For the referred patients, this database will contain information related to the following:

* Past medical history
* Obesity-related Medical co-morbidities (HTN, hyperlipidemia, e.g.)
* Lab values (fasting lipids, glucose, LFTs, HbA1c)
* Anthropometric data (ht, weight, BMI) and select vital signs (BP, HR)
* Fitness testing data
* Demographic data (age, gender, ethnicity, socioeconomic status, geographical address)
* Answers to a lifestyle, attitudes, and health habits survey
* Answers to a program survey
* Contact information for follow up

For participating family members (parents, grandparents, siblings, e.g.) this data base will contain information related to the following:

* Past medical history
* Obesity-related Medical co-morbidities (HTN, hyperlipidemia, e.g.)
* Anthropometric data (ht, weight, BMI) and select vital signs (BP, HR)
* Demographic data (age, gender, ethnicity, socioeconomic status, geographical address)
* Answers to a lifestyle, attitudes, and health habits survey
* Answers to a program survey
* Contact information for follow up

Once the database is created a retrospective chart review will be done to collect data on patients that have completed the program. This information will be obtained from facility records and program records. Individuals who previously completed the program will be contacted and asked to provide consent to be included in the database. Only data from individuals who provide consent will be included in the database.

Participants in the program will be asked to provide consent when they enroll in the program or when they come for a follow up visit. Only data from individuals who provide consent will be included in the database.

Subjects will be followed to collect information on lifestyle maintenance and long term health outcomes.

The database will be queried regularly to provide information about the participants and program.

Descriptive statistics will be calculated to describe the study population pre and post program. Outcomes will be analyzed using appropriate statistical tests. Exploratory analysis will be conducted to detect trends.

Data will be stored in a secure location with limited access. All paper documents will be stored in a locked office in a locked cabinet. Electronic data will be stored on a limited access computer. The database will be password protected and encrypted.

All participants will be assigned a study ID number. The study ID will be used for transmission of data. Data collection forms will use the assigned study ID. All data that needs to be transmitted will be de-identified to the extent possible, password protected, and encrypted.

ELIGIBILITY:
Inclusion Criteria:

* current or past participant in the NEW Keiki program
* participating family member
* able to understand English

Exclusion Criteria:

* do not meet inclusion criteria

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be participants or family members of participants in the NEW Keiki program.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2014-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Composite measure of improvement in participant/family health to include change in Body Mass Index, Weight, Blood Pressure, Lab Values | minimum 1 year
  Change in body mass index (BMI),change in weight, change in blood pressure (BP), change in lab values
Composite measure of improvement in participant/family health to include change in lifestyle survey | minimum 1 year
  Change in lifestyle survey about diet/nutrition and behaviors
Composite measure of improvement in participant/family health to include change in fitness testing data | minimum 1 year
  Change in fitness testing data

CONTACTS AND LOCATIONS:
Overall Officials: Malia Shimokawa, MD, Principal Investigator — Kapiolani Medical Center For Women & Children
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States